CLINICAL TRIAL: NCT06580015
Title: Posluma (18F-rhPSMA) PET Guided Radiotherapy Planning in Prostate Cancer: A Prospective Study Evaluating POSLUMA PET Tumor Detection on Radiation Therapy Planning and on BGRT Planning on the RefleXion X1 System
Brief Title: [18F]-rhPSMA PET-CT Imaging Performance in Patients With Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 24163; NCI-2024-06849 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24163 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-08-23; First posted 2024-08-30 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device Feasibility ([18F]-rhPSMA PET-CT, X1 RMRS PET-CT) (Experimental): Patients receive SOC flotufolastat F-18 gallium IV and undergo PET-CT on study. Patients then undergo X1 RMRS PET-CT imaging-only session 120 minutes post-injection.
  Interventions: Procedure: Computed Tomography; Other: Flotufolastat F-18 Gallium; Other: Medical Device Usage and Evaluation; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET-CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Flotufolastat F-18 Gallium — Given IV
  Other Names: (18F)-rhPSMA-7.3; 18F-rhPSMA-7.3; 18FrhPSMA-7.3; F-18-rhPSMA-7.3; Fluorine F 18 Radiohybrid PSMA-7.3; Fluorine F 18 rhPSMA-7.3; Fluorine-18 rhPSMA-7.3; Posluma; rhPSMA-7.3 (18F)
Other: Medical Device Usage and Evaluation — Undergo X1 RMRS PET-CT
Procedure: Positron Emission Tomography — Undergo PET-CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This clinical trial evaluates [18F]-rh PSMA positron emission tomography (PET)-computed tomography (CT) imaging performance in patients with prostate cancer. PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of tracer, in the case of this research, 18F-rhPSMA. Because some cancers take up [18F]-rhPSMA, cancer cells can be seen with PET. CT utilizes x-rays that traverse body from the outside. CT images provide an exact outline of organs and potential inflammatory tissue where it occurs in patient's body. Posluma (18F-rhPSMA) is an approved prostate-specific membrane antigen (PSMA) imaging agent for prostate cancer. The RefleXion Medical Radiotherapy System (RMRS) is designed to facilitate delivery of biology-guided radiotherapy (BgRT). The system uses PET emissions to guide radiotherapy delivery in real-time and has been studied for use with fludeoxyglucose (FDG) (which is an agent used in standard PET-CT scans that targets glucose). Information gathered from this study may help researchers to improve PET-CT imaging on the RefleXion system. This information will be used in the future to improve planning and delivery of radiation therapy that will target (in real time) the signal released from the [18F]-rhPSMA PET-CT tracer. Comparing the imaging from the standard of care [18F]-rh PSMA PET-CT with the imaging from RMRS may help improve the quality of the imaging captured on the RMRS for detection of imaging signals in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the imaging performance of flotufolastat F-18 gallium ([18F]-rhPSMA) PET-CT imaging subsystem of the RefleXion Medical Radiotherapy System Device in patients with lesions detected on standard-of-care (SOC) [18F]-rhPSMA PET-CT on the same day.

SECONDARY OBJECTIVES:

I. To evaluate the frequency that SOC Posluma imaging will result in the ability to distinctly identify and separate PET activity from bladder activity to aid in the detection, lesion contouring, RT planning and RT delivery for intra-prostatic lesions, prostate bed lesions (salvage RT) or lesions near the bladder.

II. To evaluate the frequency that SOC Posluma imaging will result in a change in radiotherapy planning through either exclusion due to extra-pelvic metastatic disease or detection of disease that results in a modification of RT field coverage or dose.

III. Evaluate the potential for using the X1 RMRS PET used to generate an acceptable BgRT plan such that dosimetric parameters for the target and the nearby normal anatomy are met based on investigator assessment.

OUTLINE:

Patients receive SOC flotufolastat F-18 gallium intravenously (IV) and undergo PET-CT on study. Patients then undergo X1 RMRS PET-CT imaging-only session 120 minutes post-injection.

After completion of study intervention, patients are followed up within 72 hours of PET imaging-only session.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age: ≥ 21 years
* Patients with SOC [18F]-RhPSMA PET-CT in whom a PET avid lesion is identified
* Able to get same day X1 RMRS PET

Exclusion Criteria:

* Known psychiatric or substance abuse disorder that would interfere with conduct of the study
* Patient weight exceeding the weight limit (450 pounds) outlined per X1 RMRS specifications sheet

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-01-09 (Estimated); Study Completion 2027-01-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of imaging performance of the [18F]-rhPSMA positron emission tomography (PET)-computed tomography (CT) on the X1 RefleXion Medical Radiotherapy System (RMRS) | Up to 72 hours after completion of imagining session
  Will compare the performance of the [18F]-RhPSMA PET-CT subsystem on the RefleXion X1 system to detect selected lesions in patients with prostate cancer with the SOC diagnostic [18F]- RhPSMA PET-CT. One key metric will be the percent of patients with lesions identified on SOC PET-CT that are not identified on X1 (false negatives if considering SOC the true standard). With 25 patients with lesions detected by SOC Posluma PET who undergo X1 scanning, there is at least 93% chance of finding a false negative on X1 if the true false negative rate is 10%. With 25 patients, if there are no false negatives, a false negative rate of 11.3% or above can be ruled out with a type I error <5%. Any discordances will be documented, and the final disposition recorded after a discussion between the radiation oncologist and the nuclear medicine radiologist. Graphical presentations will be provided to compare SOC positive lesions and X1 positive lesions, and SOC positive lesions and X1 neg

SECONDARY OUTCOMES:
Incidence of change in treatment planning based on SOC Posluma | Up to 72 hours after imaging session
  Will be assessed in a descriptive manner.
Percent of cases where X1 RMRS PET data can be used to generate an acceptable biology-guided radiotherapy (BgRT) plan | Up to 72 hours after imaging session
  The true positive lesions identified on the X1 PET images will be identified and used for BgRT planning. Simulated planning using the RefleXion treatment planning software will be performed, and the radiation dose to organs at risk calculated. Principal investigator will determine whether this plan is acceptable or not. The percent of cases in which RefleXion [18F]-RhPSMAcPET data led to an acceptable plan will be recorded (descriptive statistics). Descriptive statistics will be utilized to quantify results. Mean, standard deviation, IQR, and range will be reported for each continuous variable. Frequency and percentage will be reported for categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y Wong, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States